CLINICAL TRIAL: NCT07075965
Title: Calcium Channel Blocker in Myotonic Dystrophy Type 1 (CAP DM1)
Brief Title: Calcium Channel Blocker in Myotonic Dystrophy Type 1
Acronym: CAP DM1
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Johanna Hamel, Associate Professor - Department of Neurology, NMD (SMD), University of Rochester
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00010646
Record Dates: First submitted 2025-07-10; First posted 2025-07-20 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Myotonic Dystrophy 1
MeSH Terms: conditions — Myotonic Dystrophy | interventions — Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort A (Experimental): Amlodipine 5 mg
  Interventions: Drug: Amlodipine
- Cohort B (Experimental): Amlodipine 10 mg
  Interventions: Drug: Amlodipine

INTERVENTIONS:
Drug: Amlodipine — Evaluating 2 different doses of amlodipine, after an initial titration phase (2.5 mg daily), amlodipine is increased to the target doses of 5 mg and 10 mg

SUMMARY:
This is a Phase 1 clinical trial designed to evaluate the safety and tolerability of amlodipine, a calcium channel blocker, in adults with Myotonic Dystrophy Type 1 (DM1). Amlodipine is being studied to see if it can improve muscle strength, reduce stiffness (myotonia), and improve function by modifying calcium flow in muscle cells. All participants will receive amlodipine starting at 2.5 mg daily for 2 weeks, then 5 mg for 4 weeks. After that, participants will be randomly assigned to continue on 5 mg or increase to 10 mg for an additional 4 weeks. The main goals are to assess changes in blood pressure and any adverse events to determine whether the drug is safe in this population. The study will also explore how amlodipine affects muscle strength, mobility, fatigue, and daily function using clinical tests and questionnaires. Findings will inform a future phase 2 trial.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female between the ages 18 and 65, inclusive.
* A genetically confirmed diagnosis of DM1, having a repeat expansion in the DMPK gene with at least 100 CTG repeats.
* Grip strength less than 50% predicted based on age, height, and sex.
* Video hand opening time is 4 sec or greater for at least one hand.
* Ambulatory and able to walk 10 meters.
* Willingness to discontinue anti-myotonia drugs at least 2 weeks prior to screening.
* Highly effective method of contraception in women with childbearing potential.

Exclusion Criteria:

* Congenital DM1 as defined by symptom onset in the first 4 weeks of life.
* Abnormal liver function tests (LFTs): alanine aminotransferase (ALT), or aspartate aminotransferase (AST) >3 x upper limit of normal. Total bilirubin > 1.5 mg/dL, or INR > 1.3, or evidence of current active or chronic infection with hepatitis C, hepatitis B or other hepatobiliary conditions other than DM1 (or attributed to DM1) that cause abnormal liver laboratory parameters (e.g., hemochromatosis, Wilson's disease, autoimmune hepatitis)
* Current or recent infection requiring antibiotic treatment within 2 weeks prior to screening.
* Abnormal vital signs, including systolic blood pressure < 90 mmHg and diastolic blood pressure < 60 mmHg.
* Treatment with concomitant medications with potential interactions with amlodipine, these may include but are not limited to sildenafil, cyclosporin, atorvastatin at high dosages (80 mg daily), simvastatin (at dosages higher than 20 mg daily) or strong inhibitors of CYP3A4.
* A history of syncope.
* A history of symptomatic hypotension.
* Initiation or change in doses of concomitant medications, including herbal supplements, if in the opinion of the Investigator, may impact the results of the study.
* Women of childbearing potential must have a negative pregnancy test, cannot be planning a pregnancy, and cannot be breastfeeding at any time during the study.
* Known history of substance and/or alcohol abuse within one year prior to screening.
* The presence of comorbidities that, in the opinion of the Investigator, may influence study results, including, but not limited to, uncontrolled diabetes, generalized or mononeuropathy of the upper extremities, or cervical radiculopathy resulting in weakness and atrophy.
* Concurrent treatment with calcium channel blocker.
* Known ischemic or non-ischemic moderate or severe heart failure as defined by symptoms suggestive of heart failure or reduced left ventricular ejection fraction (LVEF) on echocardiogram < 55%.
* Moderate or severe aortic stenosis or other obstruction of the left ventricle outflow tract.
* Known sensitivity or allergy to amlodipine.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-12-07 (Estimated); Primary Completion 2030-10-01 (Estimated); Study Completion 2030-10-01 (Estimated)

PRIMARY OUTCOMES:
Number of Subjects Who Provided Informed Consent | Baseline
  The total number of participants who signed the informed consent document and were enrolled in the study.
Number of Completed Study Visits | Baseline to End of Study at week 10
  The total number of completed study visits, averaged across all enrolled participants. A visit is considered completed if all required procedures for that visit were performed.
Number of Subjects Who Completed the Study Without Drug Discontinuation | Baseline to End of Study at week 10
  Number of participants who completed all study visits and remained on study drug throughout the study period without permanent discontinuation due to adverse events, withdrawal, or protocol deviations.
Number of Subjects Who Completed the Study | Baseline to End of Study at week 10
  Number of participants who completed all required study visits and procedures through the final study visit.

SECONDARY OUTCOMES:
Mean Change in Systolic Blood Pressure | Baseline to End of Study at week 10
  Systolic blood pressure (SBP) will be measured using a standardized automated sphygmomanometer in a seated position after 5 minutes of rest. The mean change will be calculated as the difference between SBP at the final study visit and baseline
Number of Participants With Non-Serious Adverse Events | Baseline to End of Study at week 10
  Number of participants who experienced at least one non-serious adverse event, as determined by investigator assessment and participant report. Events will be recorded according to MedDRA coding guidelines.

IPD SHARING:
Plan to Share IPD: No